CLINICAL TRIAL: NCT02762721
Title: Molecular Analysis of Oncogenes in Tumor Samples From Adult Patients With Intrahepatic Cholangiocarcinoma or Mixed Hepatocellular-Cholangiocarcinoma
Brief Title: Analysis of Oncogenes in Intrahepatic Cholangiocarcinoma or Mixed Hepatocellular-Cholangiocarcinoma in Tumor Tissue Samples
Status: Completed | Type: Observational
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Other Study IDs: ARQ NIS-001
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Intrahepatic Cholangiocarcinoma; Mixed Hepatocellular Cholangiocarcinoma; Cholangiocarcinoma
Keywords: FGFR2 fusion; iCCA; mixed HCC-CCA; Intrahepatic Cholangiocarcinoma; Mixed Hepatocellular Cholangiocarcinoma; Cholangiocarcinoma; ArQule
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A minimum of 1 cubic mm of tumor tissue (archival) with at least 50% nucleated tumor cell content is required.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to estimate the frequency of FGFR2 fusions in archived intrahepatic cholangiocarcinoma (iCCA) or mixed hepatocellular-cholangiocarcinoma (HCC-CCA) tumor samples

DETAILED DESCRIPTION:
This is a non-interventional, observational study of archived human tissue samples; no surgical procedures will be required and no treatment will be provided as part of this study. Approximately 150 archived tissue samples obtained from patients with iCCA or mixed HCC-CCA will be analyzed for somatic alteration status and will include cholangiocarcinoma-specific FGFR2 fusion isoforms.

ELIGIBILITY:
Inclusion Criteria:

* If required by law or local regulations (i.e., the sample is from an identifiable subject), signed written informed consent should be granted prior to use of the sample in the study
* ≥ 18 years of age
* Histologically or cytologically confirmed iCCA or mixed HCC-CCA, who are/were eligible for systemic therapy (samples collected prior to initiation of the systemic therapy may be submitted for testing)
* Have one or more formalin fixed and paraffin embedded blocks available. If blocks are not evaluable, 7-10 unstained, non-baked slides with 5-micron thick sections with at least 20% tumor tissue should be available. (Potential participants who are scheduled to undergo surgical treatment may agree to provide surplus of tissues not required for diagnosis and have to provide informed consent prior to the surgery.)

Exclusion Criteria:

* Not applicable: Patients must meet all of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and fifty archived tumor tissue samples from patients with iCCA or mixed HCC-CCA will be collected from five to fifteen research sites in the United States and Italy and/or from commercially available sources. No new surgical procedures will be required and no treatment will be provided as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Estimate the frequency of FGFR2 fusions in archived iCCA or mixed HCC-CCA tumor tissue samples | Archived tumor samples will be collected through study completion, up to 18 months
  Archived tumor samples will be collected and analyzed using a Next Generation Sequencing panel.

SECONDARY OUTCOMES:
Determine the frequency of potential actionable mutations or genetic alterations in iCCA or mixed HCC-CCA | Archived tumor samples will be collected through study completion, up to 18 months
  Archived tumor samples will be collected and analyzed using a Next Generation Sequencing panel.
Formulate genetic screening recommendations for newly diagnosed patients with iCCA or mixed HCC-CCA | Archived tumor samples will be collected through study completion, up to 18 months
  Archived tumor samples will be collected and analyzed using a Next Generation Sequencing panel.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Atlanta, Georgia
  - Seattle, Washington
- Italy (4):
  - Rozzano, MI
  - Benevento
  - Milan
  - Pisa